CLINICAL TRIAL: NCT04066075
Title: Beacon Sensors & Telerehabilitation to Assess & Improve Use of Devices for Visual Functioning
Brief Title: Beacon Sensors and Telerehabilitation for Low Vision
Acronym: BeST-AID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Eye Institute (NEI) (NIH); American Academy of Optometry (Other); Southern California College of Optometry at Marshall B. Ketchum University (Other); New England College of Optometry (Other); University of Nebraska (Other); Mid Michigan Health Centers (Other); Eye Vision Associates (Unknown); See What You Miss Optometry (Unknown); Low Vision Services, PLC (Unknown); Pacific Vision Foundation (Other); Boston University (Other)
Responsible Party: Principal Investigator, Ava K. Bittner, OD, PhD, Associate Professor of Ophthalmology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #19-000267 and #18-002041
Record Dates: First submitted 2019-08-19; First posted 2019-08-26 (Actual); Results first posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Low Vision
MeSH Terms: conditions — Vision, Low

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Telerehabilitation with low vision provider (Experimental)
  Interventions: Behavioral: Low Vision Rehabilitation
- Telerehabilitation w/ low vision provider plus tele-extender (Experimental)
  Interventions: Behavioral: Low Vision Rehabilitation
- Usual Care (active control) (Active Comparator)
  Interventions: Behavioral: Low Vision Rehabilitation

INTERVENTIONS:
Behavioral: Low Vision Rehabilitation — Low Vision Rehabilitation for use of magnification devices for near reading tasks

SUMMARY:
The successful application of magnification devices for reading and daily tasks is predicated on their correct use by individuals with low vision (LV). Barriers related to transportation, geography, and/or co-morbidities often limit LV patients' ability to attend several in-office training sessions as part of low vision rehabilitation (LVR) to optimize visual function with magnification devices. A promising solution is real-time videoconferencing to provide telerehabilitation, involving remotely delivered LVR services by a LVR provider in office to a patient at home. Telerehabilitation for LV appears to be feasible and acceptable by both patients and LVR providers, yet there are no published outcomes on the potential to improve patients' visual functioning. Another key issue in LVR is the need for an effective system to continually assess how patients are functioning at home. Ideally this would involve a non-invasive, efficient method to assess when magnifier device abandonment occurs, so that a timely telerehabilitation session can be initiated. Small Bluetooth low energy beacon sensors attached to the handles of magnifiers can collect real-time data regarding minute-to-minute environmental changes, which might serve as an indicator of magnifier use by LV patients at home. Specifically, the investigators propose to assess the potential for telerehabilitation to enhance visual function by providing remotely-delivered LVR training to use magnification devices. Following one in-office training session for new magnification device(s), the investigators aim to determine if there is additional gain in visual functioning by randomizing subjects to telerehabilitation or additional in-office LVR (active control). Participants will be assessed before and after two consecutive periods: (1) one month after a single LVR training session, followed by (2) up to three LVR sessions over a three month period either via telerehabilitation in the participants' homes or LVR in-office. The investigators will determine which patient characteristics and/or magnification devices are most likely to benefit from telerehabilitation. The investigators will also determine whether data from Bluetooth beacon sensors are valid indicators of hand-held magnifier device usage by LV patients at home. The study investigators will deploy Estimote Sticker beacon sensors to subjects randomized to telerehabilitation or additional in-office LVR during the same study period. It is anticipated that beacon sensors will measure significantly increased temperature and/or motion when placed on the part of the magnification device held by LV patients while performing daily activities. Beacon sensor data will determine if it is feasible to assess when magnification devices are used, and if the frequency of magnifier use changes following telerehabilitation or in-office LVR. This work will evaluate and refine the procedures for implementing these technologies for LVR, in order to develop future randomized controlled trial protocols. The investigators envision that telerehabilitation and beacon sensors could improve LV patient outcomes by providing follow-up LVR services in a more efficient and timely manner.

ELIGIBILITY:
Inclusion Criteria:

* Any level of vision loss due to any ocular disease who are age 18 and older, and who have received new magnification device(s) for the first time (i.e., hand-held optical magnifiers, portable electronic video magnifiers, some stand magnifiers and CCTVs) from one of our participating sites.

Exclusion Criteria:

* schedules not permitting participation in planned study visits (including planning to move or take extended vacation during study period),
* inability to understand study procedures or communicate responses to visual stimuli in a consistent manner (cognitive impairment as per TICS),
* substance abuse,
* significant hearing loss (unable to hear communication by phone or via videoconferencing),
* significant medical condition likely to limit participation or lifespan, individuals who require other types of LVR training or intervention (e.g., technology/computer skills, psychosocial),
* magnifier device has features that would not work in conjunction with the beacon sensors: (1) hands-free and do not have a place where the patient's hand is holding the device during use (therefore, they would not register a significant change in temperature), and/or (2) no surface area of at least 1"x1" to which the beacon sensor could be attached without interfering with the device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ava K Bittner, OD, PhD, Principal Investigator — UCLA Stein Eye Institute
Locations (11):
- United States (11):
  - Southern Califonia College of Optometry, Fullerton, California
  - Chan Family Optometry, Grass Valley, California
  - UCLA Stein Eye Institute, Los Angeles, California
  - Frank Stein & Paul S. May Center for Low Vision Rehabilitation at The Eye Institute, San Francisco, California
  - See What You Miss Optometry, Santa Monica, California
  - New England College of Optometry, Boston, Massachusetts
  - Boston University Eye Associates, Inc., Brockton, Massachusetts
  - Mid-Michigan Eye Care, Midland, Michigan
  - University of Nebraska: Weigel Williamson Center for Visual Rehabilitation at the Truhlsen Eye Institute, Omaha, Nebraska
  - Eye Vision Associates, Nesconset, New York
  - Low Vision Services, PLC: Low Vision Learning Center, Alexandria, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bittner AK, Yoshinaga P, Bowers A, Shepherd JD, Succar T, Ross NC. Feasibility of Telerehabilitation for Low Vision: Satisfaction Ratings by Providers and Patients. Optom Vis Sci. 2018 Sep;95(9):865-872. doi: 10.1097/OPX.0000000000001260. PMID 30169361
- [Background] Bittner AK, Jacobson AJ, Khan R. Feasibility of Using Bluetooth Low Energy Beacon Sensors to Detect Magnifier Usage by Low Vision Patients. Optom Vis Sci. 2018 Sep;95(9):844-851. doi: 10.1097/OPX.0000000000001266. PMID 30169359
- [Background] Bittner AK, Yoshinaga PD, Rittiphairoj T, Li T. Telerehabilitation for people with low vision. Cochrane Database Syst Rev. 2023 Jan 13;1(1):CD011019. doi: 10.1002/14651858.CD011019.pub4. PMID 36637057
- [Result] Bittner AK, Yoshinaga PD, Shepherd JD, Kaminski JE, Malkin AG, Chun MW, Chan TL, Deemer AD, Ross NC; BeST-AID Study Team. Acceptability of Telerehabilitation for Magnification Devices for the Visually Impaired Using Various Approaches to Facilitate Accessibility. Transl Vis Sci Technol. 2022 Aug 1;11(8):4. doi: 10.1167/tvst.11.8.4. PMID 35917136
- [Result] Bittner AK, Estabrook M, Dennis N. Bluetooth Low Energy Beacon Sensors to Document Handheld Magnifier Use at Home by People with Low Vision. Sensors (Basel). 2021 Oct 25;21(21):7065. doi: 10.3390/s21217065. PMID 34770374
- [Result] Kaminski JE, Yoshinaga PD, Chun MW, Yu M, Shepherd JD, Chan TL, Deemer A, Bittner AK; BeST-AID Study Team. Value of Handheld Optical Illuminated Magnifiers for Sustained Silent Reading by Visually Impaired Adults. Optom Vis Sci. 2023 May 1;100(5):312-318. doi: 10.1097/OPX.0000000000002013. Epub 2023 Mar 22. PMID 36951854
- [Result] Bittner AK, Kaminski JE, Ross NC, Shepherd JD, Thoene SJ, Bui SZ, Yoshinaga PD; BeST-AID Study Team. Telerehabilitation Training to Facilitate Improved Reading Ability with New Magnification Devices for Low Vision. Optom Vis Sci. 2022 Oct 1;99(10):743-749. doi: 10.1097/OPX.0000000000001944. Epub 2022 Sep 6. PMID 36067410
- [Result] Bittner AK, Kaminski JE, Yoshinaga PD, Shepherd JD, Chan TL, Malkin AG, Deemer A, Gobeille M, Thoene SJ, Rossi A, Ross NC; BeST-AID Study Team. Outcomes of Telerehabilitation Versus In-Office Training With Magnification Devices for Low Vision: A Randomized Controlled Trial. Transl Vis Sci Technol. 2024 Jan 2;13(1):6. doi: 10.1167/tvst.13.1.6. PMID 38214688

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period occurred from October 10, 2019 through December 14, 2022 at academic medical or optometric clinical centers or private optometric practices.
Pre-assignment Details: Enrolled participants were excluded from the study before randomization assignment to arms or groups if they did not complete the baseline study assessments by phone.
Groups:
- Telerehabilitation With Low Vision Provider: Remote training for newly prescribed magnification devices via Zoom videoconferencing with the vision rehabilitation provider in-office and the participant at home. The training for magnifiers was individualized based on participants' needs, by providing verbal instructions to adjust placement of the reading material and/or magnifier, including feedback on working distance, viewing angle, movement and/or obtaining appropriate magnification levels and field of view while reading at near.
- Usual Care (Active Control): Training provided in-office or clinical settings in-person for the use of newly prescribed magnification devices that was individualized based on participants' needs. The training for magnifiers involves instructions to adjust placement of the reading material and/or magnifier, including feedback on working distance, viewing angle, movement and/or obtaining appropriate magnification levels and field of view while reading at near.
Period: Overall Study
Arm/Group | Telerehabilitation With Low Vision Provider | Usual Care (Active Control)
Started | 38 | 23
Completed | 29 | 18
Not Completed | 9 | 5
Not completed — Lost to Follow-up | 3 | 3
Not completed — no longer eligible or technical issue with intervention or data | 4 | 0
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Population: Participants were not included in the analysis if they were lost to follow-up (n=6), discontinued the telerehabilitation intervention due to technical issues (n=1), discontinued the trial since they were too busy (n=3) or no longer interested (n=1), became no longer eligible per inclusion/exclusion criteria (n=2), or did not have completed study assessment at 1-month or 4-months (n=3).
Groups:
- Total: Total of all reporting groups
Arm/Group | Telerehabilitation With Low Vision Provider | Usual Care (Active Control) | Total
Number analyzed (Participants) | 38 | 23 | 61
Age, Continuous [Median (Full Range); unit: years] | 70 [20 to 93] | 72 [25 to 91] | 71 [20 to 93]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants were not included in the analysis if they were lost to follow-up (n=6), discontinued the telerehabilitation intervention due to technical issues (n=1), discontinued the trial since they were too busy (n=3) or no longer interested (n=1), became no longer eligible per inclusion/exclusion criteria (n=2), or did not have completed study assessment at 1-month or 4-months (n=3).
  Participants
    number analyzed (Participants) | 29 | 18 | 47
    Female | 20 | 11 | 31
    Male | 9 | 7 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Participants were not included in the analysis if they were lost to follow-up (n=6), discontinued the telerehabilitation intervention due to technical issues (n=1), discontinued the trial since they were too busy (n=3) or no longer interested (n=1), became no longer eligible per inclusion/exclusion criteria (n=2), or did not have completed study assessment at 1-month or 4-months (n=3).
  Participants
    number analyzed (Participants) | 29 | 18 | 47
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 4 | 2 | 6
    White | 23 | 14 | 37
    More than one race | 2 | 0 | 2
    Unknown or Not Reported | 0 | 1 | 1
Activity Inventory: Reading Ability [Mean (Standard Deviation); unit: logits] — The 'Activity Inventory' is a questionnaire or patient reported outcome measure to assess reading ability during activities of daily living. Higher values represent better reading ability. Baseline scores ranged from -2.95 to 0.62. Population: Participants were not included in the analysis if they were lost to follow-up (n=6), discontinued the telerehabilitation intervention due to technical issues (n=1), discontinued the trial since they were too busy (n=3) or no longer interested (n=1), became no longer eligible per inclusion/exclusion criteria (n=2), or did not have completed study assessment at 1-month or 4-months (n=3).
  logits
    number analyzed (Participants) | 29 | 18 | 47
    (all) | -0.61 (0.88) | -0.54 (0.75) | -0.58 (0.82)
logMAR distance best-corrected visual acuity [Median (Full Range); unit: logMAR units] — Population: Participants were not included in the analysis if they were lost to follow-up (n=6), discontinued the telerehabilitation intervention due to technical issues (n=1), discontinued the trial since they were too busy (n=3) or no longer interested (n=1), became no longer eligible per inclusion/exclusion criteria (n=2), or did not have completed study assessment at 1-month or 4-months (n=3).
  logMAR units
    number analyzed (Participants) | 29 | 18 | 47
    (all) | 0.50 [0.18 to 1.5] | 0.42 [0.06 to 1.0] | 0.48 [0.06 to 1.5]
Newly Prescribed Magnifier Type [Count of Participants; unit: Participants] — Population: Participants were not included in the analysis if they were lost to follow-up (n=6), discontinued the telerehabilitation intervention due to technical issues (n=1), discontinued the trial since they were too busy (n=3) or no longer interested (n=1), became no longer eligible per inclusion/exclusion criteria (n=2), or did not have completed study assessment at 1-month or 4-months (n=3).
  Participants
    number analyzed (Participants) | 29 | 18 | 47
    hand-held optical LED magnifiers | 20 | 13 | 33
    stand optical LED magnifier | 3 | 3 | 6
    Portable electronic magnifier | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Activity Inventory
Description: change in the 'Activity Inventory' questionnaire; scores for reading ability were Rasch analyzed in logit units with higher or positive scores indicating less difficulty (i.e., improvement)(Higher values represent a better outcome/ability). Range of changes from 1 month to 4 months after receiving a magnification device were -2.06 to 2.59.
Time Frame: change from 1 month to 4 months after receiving a magnification device
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: logit
Arm/Group | Telerehabilitation With Low Vision Provider | Usual Care (Active Control)
Number analyzed (Participants) | 29 | 18
logit | 0.44 [0.08 to 0.80] | 0.43 [0.15 to 0.71]
Statistical Analysis 1: Comparison: Telerehabilitation With Low Vision Provider vs Usual Care (Active Control); Multilevel modeling in linear regression analyses accounted for within-patient correlations for the 3 assessments at baseline, 1-month and 4-months. Rasch analysis using the method of successive dichotomizations was applied to estimate person measures. Power calculation: a matched pairs t-test revealed 18 subjects per group would detect a within-subject mean improvement of 0.14-logits with 0.17-logits standard deviation for the differences, 0.80 power and 0.05 type 1 error probability; Test type: Superiority; p = 0.73, Multilevel linear regression model — The p-value represents the difference between telerehabilitation and usual care

2. Secondary Outcome: MNread Test of Reading Acuity
Description: change in reading test measured during the telerehabilitation sessions for participants who completed the MNread at two telerehabilitation sessions to indicate their reading acuity (smallest size read in logMAR units)
Time Frame: between 1 month and 4 months
Population: Participants were not included in the analysis if they were in the usual care group, had 2 telerehabilitation sessions at which the MNRead test was administered, if they were lost to follow-up (n=6), discontinued telerehabilitation intervention due to technical issues (n=1), discontinued the trial since they were too busy (n=3) or no longer interested (n=1), became no longer eligible per inclusion/exclusion criteria (n=2), or did not have completed study assessment at 1-month or 4-months (n=3).
Measure: Mean (95% Confidence Interval); unit: acuity (logMAR)
Arm/Group | Telerehabilitation With Low Vision Provider
Number analyzed (Participants) | 14
acuity (logMAR) | 0.08 [0.001 to 0.16]

3. Secondary Outcome: Geriatric Depression Scale (GDS)
Description: change in questionnaire; scale ranges from 0 to 15 with higher values indicating greater depression
Time Frame: baseline, 4 months
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: points
Arm/Group | Telerehabilitation With Low Vision Provider | Usual Care (Active Control)
Number analyzed (Participants) | 29 | 18
points | -0.14 [-1.18 to 0.89] | 1.11 [-0.29 to 2.52]

4. Secondary Outcome: Hospital Anxiety & Depression Scale
Description: change in questionnaire; subscales range from 0 to 21 for both anxiety and depression with higher values indicating greater depression or anxiety
Time Frame: baseline, 4 months
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: points
Arm/Group | Telerehabilitation With Low Vision Provider | Usual Care (Active Control)
Number analyzed (Participants) | 29 | 18
points
  Depression | -0.29 [-1.16 to 0.59] | 0.22 [-1.04 to 1.48]
  Anxiety | -0.50 [-1.42 to 0.42] | 0.72 [-0.63 to 1.74]

5. Secondary Outcome: MNread Test of Reading Speed
Description: change in reading test measured during the telerehabilitation sessions for participants who completed the MNread at two telerehabilitation sessions to indicate their log reading speed measured as words per minute.
Time Frame: between 1 month and 4 months
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: log reading speed (log words per minute)
Arm/Group | Telerehabilitation With Low Vision Provider
Number analyzed (Participants) | 14
log reading speed (log words per minute) | 0.18 [0.06 to 0.29]

ADVERSE EVENTS:
Time Frame: from enrollment (baseline) until end of follow-up at ~4-months
Description: Adverse events were all self-reported
Arm/Group | Telerehabilitation With Low Vision Provider | Usual Care (Active Control)
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/18
Other Adverse Events (participants affected / at risk) | 0/29 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT04066075/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/75/NCT04066075/ICF_001.pdf